CLINICAL TRIAL: NCT06159413
Title: LUMBAR MULTIFIDUS MUSCLES FUNCTION AMONG PATIENTS WITH LOW BACK PAIN: VIRTUAL REALITY VERSUS STABILIZATION EXERCISES.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Mohamed Raafat Atteya, Assistant Professor, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UoH1
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain; Low Back Pain, Mechanical
Keywords: Pain
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded controlled study.
Who Masked: Participant
Masking Description: Sixty LBP participants will be divided into three groups in a 1:1:1 ratio, 20 in each group (control group, stabilizing exercises, and virtual reality rehabilitation system). All three groups received training three days per week throughout the Six-week treatment session.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: VIRTUAL REALITY — LUMBAR MULTIFIDUS MUSCLES FUNCTION AMONG PATIENTS WITH LOW BACK PAIN: VIRTUAL REALITY VERSUS STABILIZATION EXERCISES.
  Other Names: STABILIZATION EXERCISES

SUMMARY:
Abstract:

Background: The multifidus muscle, the most medially located back muscle and the largest muscle that spans the lumbosacral junction serves to provide dynamic stability to the spinal column. Virtual reality and core stabilization exercises are commonly used for balance training in musculoskeletal conditions. The knowledge regarding the effective implementation of these training protocols in patients suffering from chronic low back pain (LBP) is insufficient.

Objective: The purpose of the present study is to investigate the efficacy of virtual reality versus stabilization exercises on lumbar multifidus muscle function among patients with low back pain.

Design: Randomized, double-blinded controlled study. Participants: Sixty LBP participants will be divided into three groups in a 1:1:1 ratio, 20 in each group (control group, stabilizing exercises, and virtual reality rehabilitation system). All three groups received training three days per week throughout the Six-week treatment session.

Outcome measures: Evaluation of pain by the visual analog scale (VAS), Level of functional impairments by Oswestry Disability Index and Accuracy of lumbar repositioning measurement by Biodex system will be measured at baseline and after Six weeks.

DETAILED DESCRIPTION:
Introduction:

Low back pain (LBP) is still a significant concern for the public. Health concerns in affluent nations despite advances in our understanding of spinal illnesses. The issue is significant because of its socioeconomic and psychological implications and the shortcomings of many suggested preventive or cure measures (Almazrou et al., 2020; Schmidt et al., 2020). Up to 75% of people will experience low back discomfort at some point with some extent of functional difficulties (De Souza et al., 2019).

With its distinct stabilizing function, the multifidus muscle, which spans the lumbosacral junction and is situated medially in the back, gives the spinal column dynamic stability (Zwambag et al., 2019). It is crucial to remember that people with low back pain may have a multifidus muscle problem, which includes critical structural alterations such as atrophy and the replacement of muscular tissue with fatty infiltrates (Shahidi et al., 2017). A lack of proprioception and abnormal recruitment patterns are two further motor control deficiencies noted (Chua et al., 2022; Shahidi et al., 2023).

Several studies have linked Multifidus muscle atrophy to LBP in both acute and chronic stages (Maas et al., 2018). This muscle loss is not due to atrophy from lack of usage; multifidus activity is reflexively inhibited (Masse-Alarie et al., 2016a). Atrophy of the spinal muscles can lead to instability and recurrent back problems (Massé-Alarie et al., 2016b). Appropriate lumbosacral position sensing depends on the multifidus muscles' muscle spindles. Lower back pain (LBP) sufferers typically have a less accurate and exact sense of their position than healthy individuals. Multifidus muscle atrophy may result in muscle spindle dysfunction, which can limit muscle spindle input and impair segmental stability and spinal proprioception (Crawford et al., 2019; Gabel et al., 2021).

Computer technology, virtual reality (VR), employs sensory feedback to provide users with an experience that mimics real-life activities and events. People can improve their motor abilities in a fashion that mimics the real world by using a three-dimensional virtual environment (Park et al., 2019). Virtual reality systems are well known for their distinctive qualities of interactivity and immersion. Utilizing several sense channels, such as sight, hearing, and touch, requires interaction. The degree of interaction with the virtual environment, on the other hand, is related to immersion (Coburn et al., 2017; Papadopoulos et al., 2021). To influence the cognitive processes involved in motor control, one needs a sense of "degree of presence," or awareness of one's existence in a certain scenario. Virtual reality technology makes the development of interactive training regimens that target various muscles, joints, coordinated movements, or the complete body easier (Levac et al., 2019; Tieri et al., 2018). There is currently a dearth of research on how VR affects the function of the multifidus muscles in people with LBP.

Even though much research has been done, the best course of action for treating persistent LBP and the value of different physical therapy are still debatable. A various physical therapy methods for treating LBP have also been conducted without the superior of one technique on the others (Ahmed, Maharaj, et al., 2021; Ahmed, Nadasan, et al., 2021; Mohamed Kamel et al., 2019).

This study compares the effects of lumbar stabilizing exercises and virtual reality on the multifidus muscle's cross-sectional area, the lumbar spine's ability to accurately realign pain levels, and functional limitations in people with chronic lower back pain.

Methods.

Design of the trial

Using a computer random table method, the study divided the participants evenly among the three groups in a 1:1:1 ratio. The research will be randomized, controlled, and double-blinded. There will be 60 participants, 20 in each of the three groups (control group, stabilizing exercises, and virtual reality rehabilitation system). The Physical Therapy Department at the University of Hail in Saudi Arabia selected study participants from the Hail University Clinics. The research underwent approval from the Departmental Scientific Ethics Committee. Additionally, it adhered to the comprehensive reporting standards of the unified standards for reporting trials (CONSORT), ensuring full transparency. A physical therapist from the department evaluated to determine participant eligibility.

Participants:

Participants had to provide their consent and sign an informed consent form authorized by an ethics committee to be eligible for the study. The selection criteria comprised those between the ages of 30 and 50 who had been dealing with persistent lower back pain for more than three months and who graded their pain on a visual analog scale (VAS) as being between four and eight. A person will be not considered eligible for the study if they had severe musculoskeletal, neural, somatic, or psychiatric disorders, will be recovering from spinal surgery, will be abusing alcohol or drugs, will be taking part in other weight and balance-training programs, had deformities or other soft tissue injuries or bone fractures.

Patient participation:

Through a study information form, the researchers sent the 60 patients who will be initially chosen thorough instructions and information regarding the trial's goals, design, intervention techniques, outcome metrics, length, and potential risks and benefits.

Interventions:

With The Ethics Committee's Approval, the VRG, STG, and control groups will undergo four-week rehabilitation programs. A physiotherapist with five years of expertise and a good skill set completed the recovery process. The study excluded ten people who chose not to participate, eleven with joint problems, four who applied for surgery, and seven who reported significant pain (VAS score greater than 8).

Participants in the study utilized a device that encouraged balance exercises to strengthen their core muscles and increase their stability. They will be given one-on-one instructions while seated on how to use the virtual reality game (VRG). The participants' balance will be tested in this position, which also helped them become accustomed to the game's rules.

A shooting game will be present in the recent study. The game will be played on a display screen while participants sat on a virtual platform. Following the signs, they moved their trunks forward, backward, and left to right to control the game. Participants will be urged to move their spines as much as possible while staying within their discomfort thresholds. The actions in the game will be rated, and as they progressed in complexity, They have become increasingly challenging.

Measures of results

The outcome measures will be assessed at baseline and again Six weeks later.

1. Evaluation of pain:

   The visual analog scale (VAS) is a 10 cm line with 0 representing no pain and 10 representing the worst pain. It will be used to ask patients to rate how much pain they perceived. They will be told to draw a mark on the line where their level of pain will be.
2. Level of functional impairments

   To assess functional disability, we employed the Oswestry Disability Index. Ten multiple-choice questions about back discomfort and everyday activities are included. Each question has six potential answers and a maximum score of 5. Based on a few chosen statements, the ultimate score is determined.

   Score overall: (5 questions answill bed) x 100%.

   The degree of disability is determined using a scale from 0 to 50. The score reflects the severity of the condition, with higher scores indicating more profound impairment. Scores between 20% and 40% indicate significant disability, whereas those between 0 and 20% suggest mild disability. Scores between 40% and 60% indicate severe disability, and those between 60% and 80% indicate crippling disability. Lastly, an 80% to 100% score denotes bed rest for the patient (Fairbank & Pynsent, 2000; Monticone et al., 2012).
3. Accuracy of lumbar repositioning measurement

Knee blocks, leg pads, thigh straps, pelvic brace, lumbar pad, and force application straps will be used to position the person in the Biodex system. The head will be supported on a flexible rest while straps restrained the torso. The spinal range of motion created a neutral spinal posture at 30 degrees lumbar flexion. We asked participants to bend their backs as far as possible to determine the range of motion. For consistency, the dynamometer will be adjusted at zero degrees. Participants will be instructed to recall and replicate a 30° position in a practice trial. We ran this test thrice and calculated the mean deviation each time (Wilson & Granata, 2003).

Statistic evaluation

We used Levene's test to measure the participant's demographics to confirm the study's consistency. We showed the mean and standard deviation for the outcome data. We used SPSS software to conduct repeated measures and one-way ANOVA tests to determine significant changes within groups, with a statistical significance level of P 0.05. (IBM SPSS Statistics, V 23).

ELIGIBILITY:
Inclusion Criteria:

* Patients with low back pain.

Exclusion Criteria:

* Patients with pain more than 8 according to VAS.
* Any joint problems.
* Any surgical intervention.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain | 6 weeks
  The visual analog scale (VAS) is a 10 cm line with 0 representing no pain and 10 representing the worst pain. It will be used to ask patients to rate how much pain they perceived. They will be told to draw a mark on the line where their level of pain will be.
Level of functional impairments | 6 weeks
  To assess functional disability, we employed the Oswestry Disability Index. Ten multiple-choice questions about back discomfort and everyday activities are included. Each question has six potential answers and a maximum score of 5. Based on a few chosen statements, the ultimate score is determined.
Accuracy of lumbar repositioning measurement | 6 weeks
  Knee blocks, leg pads, thigh straps, pelvic brace, lumbar pad, and force application straps will be used to position the person in the Biodex system. The head will be supported on a flexible rest while straps restrained the torso. The spinal range of motion created a neutral spinal posture at 30 degrees lumbar flexion. We asked participants to bend their backs as far as possible to determine the range of motion. For consistency, the dynamometer will be adjusted at zero degrees. Participants will be instructed to recall and replicate a 30° position in a practice trial. We ran this test thrice and calculated the mean deviation each time.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed raafat Atteya, Ha'il, Ha'il Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
All data collected, including age, weight and height, will be shared